CLINICAL TRIAL: NCT02115022
Title: Endoscopic UltraSound in Potentially Resectable PAncreatic Malignancy - Does it Bear the Weight of the Rapidly Evolving Technology of Computer Tomography?
Brief Title: EUS vs. MDCT in Pancreatic Malignancy
Acronym: EUSPACT
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Colentina (Other)
Collaborators: University of Medicine and Pharmacy Craiova (Other); Iuliu Hatieganu University of Medicine and Pharmacy (Other); Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Mihai Rimbas, MD, PhD, Assistant Professor, Clinical Hospital Colentina
Other Study IDs: Col-gastro 5
Record Dates: First submitted 2014-04-13; First posted 2014-04-15 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Resectable Pancreatic Cancer
Keywords: pancreatic cancer; resectability; endosonography (EUS); multidetection computer tomography (MDCT); staging
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Potentially resectable pancreatic cancer: Patients with a confirmed pancreatic mass (suspected neoplastic) deemed resectable or borderline resectable on multislice (at least 16 simultaneously acquired slices) pancreatic protocol computed tomography (CT), fit and willing to undergo surgery with a curative (R0) intent.

SUMMARY:
Accurate staging of patients with pancreatic cancer is critical to avoid the expense, morbidity, and mortality related to unnecessary surgery. While several tests are available for assessing such patients, consensus has not been achieved on the optimal approach. As a matter of fact, pancreatic cancer staging is discussed controversially due to conflicting evidence and certainly EUS has lost grounds due to improvements in CT technology. Thus, the role of EUS and EUS-guided FNA varies among treatment centers.

The present study is designed to better define the role of EUS in predicting resectability, as compared to high resolution cross-sectional imaging.

DETAILED DESCRIPTION:
Registry procedures:

* HIGH-RESOLUTION PANCREATIC PROTOCOL COMPUTED TOMOGRAPHY (CT) SCAN EXAMINATION: performed on at least 16-section multi-detector row (MD) CT and reviewed using multi-planar reconstructions, with images obtained following the oral administration of water and pancreatic protocol intravenous iopamidol, with images acquired in the pancreatic and portal venous phases of contrast enhancement, reconstructed as thin slice (at 1 mm - pancreatic phase or 2 mm - portal venous phase increments).
* EUS EXAMINATION: performed within 2 weeks of the MDCT, aiming visualization of the pancreas, main surrounding vascular structures, celiac and mediastinal lymph nodes, liver and left adrenal gland, with EUS-FNA performed at the discretion of the investigator/examiner to confirm/exclude metastases and for the confirmation of malignancy in the primary tumor. Patients confirmed by EUS as having distant metastases are to be deferred from the planned surgical intervention.
* SURGICAL INTERVENTION: aiming to provide curative intent (R0) resection.
* HISTOPATHOLOGICAL POSTOPERATIVE STAGING: with evaluation of loco-regional invasiveness and degree of complete surgical resection (R0/R1).
* FOLLOW-UP OF PATIENTS: with phone-calls on an every 6 month basis, for up to 2 years, retaining the following data: survival (or not), date of decease and its direct cause (if applicable), the presence of tumor recurrence (or not).

ELIGIBILITY:
Inclusion Criteria:

* adult (≥ 18 years of age) patients;
* the presence of a confirmed pancreatic mass (suspected neoplastic) deemed resectable or borderline resectable on multislice (at least 16 simultaneously acquired slices) pancreatic protocol computed tomography (CT);
* patients fit and willing to undergo surgery with a curative (R0) intent;
* sign of the informed consent.

Exclusion Criteria:

* the presence of significant co-morbidities that contraindicate pancreatic resection;
* previous neo-adjuvant oncologic therapy;
* distant metastases;
* lack of discernment;
* refusal to sign the informed consent..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a confirmed pancreatic mass (suspected neoplastic) deemed resectable or borderline resectable on multislice (at least 16 simultaneously acquired slices) pancreatic protocol computed tomography (CT), fit and willing to undergo surgery with a curative (R0) intent.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Staging capability of each study procedure | Up to 2 weeks, depending on the time of the surgical intervention
  Each imaging test (MDCT and EUS) and findings at or after surgery are to be judged on their ability to provide descriptions of the primary tumor's size, location, relationship to vessels - using the terms abutment (≤180º of contact) and encasement (>180º of contact), vessel occlusion, variant vascular anatomy, a grade regarding local tumor resectability (resectable, borderline resectable, or locally advanced; R0 or R1 resection), and extent and location of extrapancreatic disease.

SECONDARY OUTCOMES:
Side-effects related to the EUS examination | Monitored for 24 hours after EUS
  Each patient will be monitored for 24 hours after the EUS examination to identify possible early complications of the procedure
Patient survival time, and tumor recurrence-free survival | Up to 2 years
  Each patient is going to be followed-up for up to 2 years after the surgical intervention an an every-6 month basis, in order to identify events such as death or tumor recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Rimbas, MD, PhD, Principal Investigator — Clinical Hospital Colentina, Carol Davila University of Medicine and Pharmacy; Cristian R Baicus, Professor, Study Chair — Clinical Hospital Colentina, Carol Davila University of Medicine and Pharmacy; Adrian Saftoiu, Professor, Study Director — Craiova research Center in Gastroenterology and Hepatology, Craiova University of Medicine and Pharmacy
Locations (5):
- Romania (5):
  - Research Center in Gastroenterogy and Hepatology, Craiova, Dolj
  - University Military Hospital, Bucharest
  - Gastroenterology Department, Clinical Hospital Colentina, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Iuliu Hatieganu University of Medicine, Cluj-Napoca